CLINICAL TRIAL: NCT05051722
Title: Leveraging Methylated DNA Markers (MDMs) in the Detection of Endometrial Cancer, Ovarian Cancer, and Cervical Cancer: a Phase II Clinical Study
Brief Title: Leveraging Methylated DNA Markers (MDMs) in the Detection of Endometrial Cancer, Ovarian Cancer, and Cervical Cancer
Acronym: ECHO
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-012833; NCI-2022-10826 (Registry Identifier: NCI)
Record Dates: First submitted 2021-09-11; First posted 2021-09-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer; Cervical Cancer; Atypical Endometrial Hyperplasia; Cervical Dysplasia; Adnexal Mass; Ovarian Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Cervical Neoplasms; Endometrial Hyperplasia; Uterine Cervical Dysplasia; Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A sample of the vaginal fluid will be collected from each study participant prior to any clinical exams or procedures.
  * A peripheral blood sample will be collected from each study participant prior to any clinical exams or procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Cohort 1 - AUB / PMB: Patients ≥45 years of age, presenting with abnormal uterine bleeding (AUB) or post-menopausal bleeding (PMB). Patients ages 18 - 44 years of age, presenting with abnormal uterine bleeding (AUB) and a risk factor for endometrial cancer (BMI ≥30 or PCOS or Tamoxifen use). These presenting symptoms clinically warrant evaluation such as an endometrial biopsy to assess for underlying endometrial cancer, endometrial hyperplasia or other endometrial pathology.
  Interventions: Diagnostic Test: Vaginal Fluid Collection; Diagnostic Test: Blood Collection
- Cohort 2 - Biopsy-proven EC or AEH or EIN: Patients ≥18 years of age with biopsy-proven endometrial cancer (EC), atypical endometrial hyperplasia (AEH), or endometrial intraepithelial neoplasia (EIN) presenting for surgical management of their endometrial pathology.
  Interventions: Diagnostic Test: Vaginal Fluid Collection; Diagnostic Test: Blood Collection
- Cohort 3 - Cervix pathology: Patients ≥18 years of age presenting for a clinically indicated colposcopy, cervical biopsy, or surgical excision, as follow-up for an abnormal Pap test or cervical mass identified on physical exam. Final clinical diagnoses within this cohort may include mild cervical intraepithelial neoplasia (CIN 1), moderate and/or severe CIN (CIN 2/3), adenocarcinoma in situ (AIS), invasive cervical cancers (adenocarcinoma or squamous cell carcinoma), or possibly benign findings.
  Interventions: Diagnostic Test: Vaginal Fluid Collection; Diagnostic Test: Blood Collection
- Cohort 4 - Benign Uterine Pathology: Patients with any of four benign gynecologic conditions including: uterine fibroids, benign endometrial polyps, adenomyosis and endometriosis. All patients enrolled in this cohort will be undergoing clinically indicated gynecologic surgery (hysterectomy, myomectomy, polypectomy, or laparoscopic tissue excision) for the specific benign gynecologic condition. Verification of the final benign diagnosis will be based on pathology diagnosis of clinically-indicated tissue removed during surgery.
  Interventions: Diagnostic Test: Vaginal Fluid Collection; Diagnostic Test: Blood Collection
- Cohort 5 - Healthy Control Women: Healthy patients with a uterus, ≥45 years of age presenting for GYN wellness exam to serve as a control group. These patients will have no clinically evident gynecologic precancers, gynecologic cancers, or clinically evident or symptomatic benign gynecologic conditions. These patients will not have known or clinically suspected AUB, PMB, fibroids, endometriosis, benign endometrial polyps, or adenomyosis, nor will they have any active gynecologic or non-gynecologic acute medical conditions.
  Interventions: Diagnostic Test: Vaginal Fluid Collection; Diagnostic Test: Blood Collection
- Cohort 6- Isolated Adnexal Mass Cohort (ovarian or fallopian mass): Patients ≥50 years of age and postmenopausal (12 months since LMP or available blood hormone levels confirming postmenopausal status) and an isolated adnexal mass or isolated bilateral adnexal masses being surgically removed. These patients may have a final diagnosis of any of the following: benign ovarian neoplasm, borderline tumor of the ovary, or clinically early-stage OC.
  Interventions: Diagnostic Test: Vaginal Fluid Collection; Diagnostic Test: Blood Collection
- Cohort 7 - OC Cohort - Biopsy proven or clinically suspected ovarian cancer (OC): Patients ≥18 years of age with ovarian cancer (OC) (clinically probable based on distribution of pelvic/abdominal masses on imaging, elevated CA-125, ascites, and/or imaging-guided biopsy proven) presenting for neoadjuvant chemotherapy or primary surgical management (debulking or staging) of their OC. The umbrella of OC also includes fallopian tube cancer and primary peritoneal cancer. All histologies are eligible for enrollment.
  Interventions: Diagnostic Test: Vaginal Fluid Collection; Diagnostic Test: Blood Collection

INTERVENTIONS:
Diagnostic Test: Vaginal Fluid Collection — A sample of vaginal fluid will be collected from each participant, prior to any exams or procedures, by a healthcare provider using a small vaginal swab.
  Other Names: Vaginal Fluid
Diagnostic Test: Blood Collection — A blood sample will be collected from each participant prior to undergoing any exams or procedures.

SUMMARY:
The overarching objective of this project is to develop a pan-gynecologic cancer detection test using gynecologic (unique endometrial, cervical, and ovarian cancer) cancer-specific methylated DNA markers and high-risk human papilloma virus (HR-HPV) detected in vaginal fluid and/or plasma.

This proposal defines Phase II MDM-based cancer detection studies in endometrial cancer (EC) and endometrial hyperplasia with atypia (AEH) in vaginal fluid and 2) ovarian cancer (OC) in plasma and vaginal fluid. Additionally, it defines necessary Phase I MDM-based cancer detection and exploratory aims to test novel cervical cancer (CC) MDMs and test the specificity of cancer-specific MDMs among various common benign gynecologic pathologies.er detection and exploratory aims to test novel cervical cancer MDMs and test the specificity of cancer-specific MDMs among various common benign gynecologic pathologies.

DETAILED DESCRIPTION:
Detection of endometrial, ovarian, and cervical cancers at an early stage vastly increases the chances of cure and may also avert morbidity secondary to surgical staging, radiation, and/or chemotherapy. Despite the great successes of cervical cancer screening, comparable early detection methods for other gynecologic cancers and their precursors are not available. While nearly 1.5 million women per year in the United States are evaluated for abnormal uterine bleeding (AUB) or postmenopausal bleeding (PMB), the most common symptom of endometrial cancer, most undergo an invasive diagnostic biopsy with the finding of benign etiology.

Vaginal bleeding is often the only presenting symptom of women ultimately diagnosed with endometrial cancer (EC) or its precursor lesion, endometrial hyperplasia(EH). More than 90% of women with EC present with vaginal bleeding. Cervical cancer and cervical dysplasia can present as intermenstrual bleeding, post-coital bleeding, or other abnormal vaginal bleeding. However, most women who present with AUB or PMB have a benign etiology.

There are approximately 70 million women ≥45 years of age in the United States based on the most recent census data. Between 4-11% of women will be worked up for perimenopausal AUB or PMB in their lifetime. As only 5-10% of those women will have an EC or EH, there is a great clinical need for a less invasive clinical diagnostic test that can reliably distinguish between benign uterine bleeding and bleeding associated with an underlying endometrial cancer, cervical cancer, or a precursor lesion.

ELIGIBILITY:
Inclusion Criteria for Cohort 1:

Patients will be ≥45 years of age and meet one of the following criteria:

* Abnormal uterine bleeding
* Postmenopausal bleeding

OR

Patients ages 18 - 44 years of age and meet these criteria

* Abnormal uterine bleeding
* One risk factor for endometrial cancer (BMI ≥30 or PCOS or Tamoxifen use)

Exclusion Criteria for Cohort 1:

* Prior hysterectomy
* Current known pregnancy diagnosis
* Any prior pelvic or vaginal radiotherapy
* Any prior cancer (except basal cell skin cancer) within the past 5 years
* Chemotherapy within the past 5 years
* Current biopsy-proven cervical, vaginal, or vulvar cancer or lower genital tract dysplasia
* Current biopsy-proven endometrial cancer or endometrial hyperplasia
* Current biopsy-proven benign endometrial polyp
* Endometrial biopsy/sampling within the preceding 1 month showing benign endometrium

Inclusion Criteria for Cohort 2:

Patients will be ≥18 years of age and meet at least one of the following criteria:

* Presence of biopsy-proven EC (any histology, including uterine carcinosarcoma) and surgical intervention planned. Surgical intervention can include any of the following: hysterectomy, D&C, hysteroscopic resection
* Biopsy showing AEH or EIN with surgical intervention planned. Surgical intervention can include any of the following: hysterectomy, D&C, hysteroscopic resection, etc)

Exclusion Criteria for Cohort 2:

* Undergoing surgical procedure for recurrent or metastatic EC
* Received preoperative neoadjuvant chemotherapy or radiotherapy for current EC diagnosis
* Prior hysterectomy
* Current known pregnancy diagnosis
* Prior or current biopsy-proven cervical cancer
* Presence of concomitant biopsy-proven cervical dysplasia
* Any prior pelvic or vaginal radiotherapy
* Any prior cancer (except basal cell skin cancer) within the past 5 years
* Chemotherapy within the past 5 years
* Prior intervention or surgery with intent to completely remove the target pathology

Inclusion Criteria for Cohort 3:

Patients will be ≥18 years of age, have a cervix and meet at least one of the following criteria:

* History of current abnormal cervical/endocervical Pap test for which the patient is presenting for colposcopy
* Cervical mass identified on physical exam and patient referred for cervical biopsy, even if colposcopy not recommended or indicated
* Planned clinically indicated surgical excisional biopsy or removal of the cervix (cold knife cone, LEEP, hysterectomy) for abnormal Pap test, cervical dysplasia, cervical mass, or biopsy-proven invasive cervical cancer (adenocarcinoma, squamous cell carcinoma, adenosquamous carcinoma, or less common primary cervical carcinomas all eligible)

Exclusion Criteria for Cohort 3:

* History of pelvic or vaginal radiotherapy
* Prior total hysterectomy (cervix removed) for any indication
* Current known pregnancy diagnosis
* Cervical mass biopsy-proven to be EC or a cancer metastatic from a non-cervical origin
* Any prior cancer (except basal cell skin cancer) within the past 5 years
* Chemotherapy within the past 5 years
* Patients presenting for colposcopy as part of lower genital tract dysplasia or cancer surveillance after prior curative intent treatment and no current Pap abnormality or cervical mass
* Prior intervention or surgery with intent to completely remove the target pathology for the current lesion / diagnosis during the current episode

Inclusion Criteria for Cohort 4:

Patients will be ≥45 years of age and should meet at least one of the following criteria:

* Undergoing hysterectomy with biopsy-proven or clinically presumed (based on imaging and/or clinical symptoms) benign gynecologic or uterine pathology of fibroids, endometriosis, adenomyosis, or benign endometrial polyps.
* Undergoing any gynecologic surgery in which a benign pathologic tissue diagnosis of fibroids, endometriosis, adenomyosis, or benign endometrial polyp is anticipated to be confirmed.

Exclusion Criteria for Cohort 4:

* Endometrial biopsy or office hysteroscopy within 2 weeks preceding the planned gynecologic surgery procedure for fibroids, endometriosis, benign endometrial polyps, or adenomyosis
* Any surgery within the past 3 months
* Prior hysterectomy
* Current known pregnancy diagnosis
* Prior or current biopsy-proven gynecologic cancer
* Current biopsy-proven AEH/EIN, cervical, vaginal, or vulvar dysplasia
* Prior pelvic or vaginal radiotherapy
* Any prior cancer (except basal cell skin cancer) within the past 5 years
* Chemotherapy within the past 5 years
* Undergoing hysterectomy for prolapse without a coexisting known or presumed benign uterine pathologic diagnosis of fibroids, endometriosis, benign endometrial polyps, or adenomyosis
* Prior intervention or surgery with intent to completely remove the target pathology for the current lesion / diagnosis during the current episode

Inclusion Criteria for Cohort 5:

Patients with a uterus will be ≥45 years of age and should meet the following criteria:

* Presenting for GYN wellness exam, ± Pap test
* No change in medical conditions, new diagnoses, or new medications within the past 6 months

Exclusion Criteria for Cohort 5:

* Pap test or cervical biopsy within the past 1 month
* Endometrial biopsy or office hysteroscopy within the past 1 month
* Any surgery within the past 3 months
* Prior hysterectomy
* Current known pregnancy diagnosis
* Prior or current biopsy-proven gynecologic cancer
* Current biopsy-proven AEH/EIN, cervical, vaginal, or vulvar dysplasia
* Prior pelvic or vaginal radiotherapy
* Any prior cancer (except basal cell skin cancer) within the past 5 years
* Chemotherapy within the past 5 years
* Criteria met for inclusion in any of the other study cohorts

Inclusion Criteria for Cohort 6:

Patients ≥50 years of age and:

* Postmenopausal
* At least 1 intact ovary
* Diagnosis of an adnexal mass or a clinical suspicion of early-stage ovarian cancer (including fallopian tube cancer)
* Planned surgery for the adnexal mass
* For vaginal fluid collection, patient must have a uterus, cervix and at least 1 intact fallopian tube* (without prior tubal ligation/occlusion)

Exclusion criteria for Cohort 6:

* Any current or prior cancer diagnosis (except basal cell or squamous cell skin cancer, non-gyn)
* Chemotherapy for cancer treatment within the past 5 years prior to collection
* Clinically suspected advanced stage ovarian cancer (Stage III or IV) on presentation, if known prior to specimen collection
* Surgical candidates for recurrent ovarian cancer
* History of pelvic or vaginal radiation therapy
* Known current synchronous endometrial cancer or hyperplasia
* Known current cervical, vaginal, or vulvar dysplasia

Inclusion criteria for Cohort 7:

Women will be ≥18 years of age and meet the following criteria:

* Presence of clinically probable ovarian, fallopian tube, or primary peritoneal cancer (all under the umbrella of OC) based on clinical findings of any/all of the following: imaging showing adnexal and/or abdominal masses consistent with probable ovarian cancer, omental caking, elevated CA125, ascites, imaging-guided biopsy consistent with OC pathology
* Newly diagnosed with ovarian, fallopian tube or primary peritoneal cancer without neoadjuvant therapy
* At least one intact ovary
* For vaginal fluid collection, patient must have a uterus, cervix and at least 1 intact fallopian tube* (without prior tubal ligation/occlusion)

Exclusion criteria for Cohort 7:

* Patients with recurrent OC
* Any current or prior cancer diagnosis (except basal cell or squamous cell skin cancer, non-gyn) within the past 5 years
* Chemotherapy for cancer treatment within the past 5 years prior to collection
* History of pelvic or vaginal radiation therapy
* Known current synchronous endometrial cancer or hyperplasia
* Known current cervical, vaginal, or vulvar dysplasia
* Current known pregnancy diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to a GYN or GYN Surgery Clinic for evaluation of symptoms or for consultation and planned procedures as outlined in the seven study cohort descriptions.
Sampling Method: Non-Probability Sample
Enrollment: 3110 (Estimated)
Dates: Start 2021-08-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Develop predictive models from a panel of EC-specific MDMs and validate their performance in identifying underlying EC and AEH within vaginal fluid in a larger, more diverse cohort. | 18 months
  Complete a phase II biomarker development study of a methylated DNA marker (MDM)-based endometrial cancer detection test performed on vaginal fluid. The phase II aspect of this biomarker development study will narrow the number of endometrial cancer MDMs within the biomarker panel in order to optimize the next phase of test development.
Develop predictive models from a panel of OC-specific MDMs and validate their performance in identifying underlying OC within vaginal fluid and plasma in a larger, more diverse cohort. | 18 months
  Complete a phase II biomarker development study of a methylated DNA marker (MDM)-based ovarian cancer detection test performed on vaginal fluid. The phase II aspect of this biomarker development study will narrow the number of ovarian cancer MDMs within the biomarker panel in order to optimize the next phase of test development.

SECONDARY OUTCOMES:
Using 95% specificity cutoffs of the final MDM EC panel, determine the false positive rate among women undergoing surgical removal of common benign gynecologic pathology | 18 months
  As part of this biomarker test development, understanding whether common non-cancerous uterine or gynecologic conditions may also lead to the finding of currently apparent endometrial cancer-specific MDMs in vaginal fluid is critical in determining specificity, positive predictive value, and negative predictive value of the test.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie N Bakkum-Gamez, M.D., Principal Investigator — Mayo Clinic
Locations (24):
- United States (24):
  - Mayo Clinic, Phoenix, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - My GYN Care, Miami, Florida
  - Genoma Research, Inc., Miami, Florida
  - Orlando Health, Orlando, Florida
  - Signature Women's Healthcare, LLC, Pembroke Pines, Florida
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Providea Health Partners, LLC, Evergreen Park, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Valley OB-GYN Clinic, Saginaw, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - The Woman's Health Pavilion, Howard Beach, New York
  - The Woman's Health Pavilion, Westbury, New York
  - Altru Health System, Grand Forks, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - Total Women's Care of the Heights, Houston, Texas
  - Medical Colleagues of Texas, LLP, Katy, Texas
  - Virginia Commonwealth University/ Massey Cancer Center, Richmond, Virginia
  - Mayo Clinic Health System - Northwest Wisconsin, Eau Claire, Wisconsin
  - Mayo Clinic Health System - Southwest Wisconsin, La Crosse, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials